CLINICAL TRIAL: NCT03873688
Title: Effects of Expiratory Muscle Training on Cough Efficacy in Children and Adolescents With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cigdem Emirza (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Sponsor-Investigator, Cigdem Emirza, Physiotherapist, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TYL-2018-31769
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Cystic Fibrosis
Keywords: expiratory muscle training; cough; respiratory muscle strength; exercise capacity
MeSH Terms: conditions — Cystic Fibrosis; Cough

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients in experimental group will perform expiratory muscle training as home programme for at least five days a week, twice a day for 15 minutes at each session during six weeks by Threshold Positive Expiratory Pressure device. The intensity of training will been setted 30% of the maximal expiratory pressure level.
  Interventions: Other: expiratory muscle training
- Sham Group (Sham Comparator): In sham group, patients will perform expiratory muscle training at home for at least five days a week, twice a day for 15 minutes at each session during six weeks by Threshold Positive Expiratory Pressure device that the intensity of training will been setted 5 cm H₂O.
  Interventions: Other: expiratory muscle training

INTERVENTIONS:
Other: expiratory muscle training — The intensity of training will been determined after assessment of maximal expiratory pressure (MEP). The first training session will perform under the supervision of a physiotherapist, patients will perform training at home. MEP measurement will reevaluate every two weeks and the intensity of training will set according to MEP levels.

SUMMARY:
Cystic fibrosis (CF) is an autosomal recessive genetic disease characterized by recurrent airway infections, affecting many systems including lung, pancreas and sweat glands. Cough is an important defense mechanism for clearing the secretions that increase in respiratory diseases. There have been studies investigating the effect of expiratory muscle training on disease groups such as chronic obstructive pulmonary disease, multiple sclerosis, parkinson's disease, and the elderly and healthy individuals. Studies that evaluating effects of expiratory muscle training in cystic fibrosis are limited in the literature. The aim of this study was to evaluate the effect of cough strength in children and adolescents with CF and the effect of expiratory muscle training program on cough strength, exercise capacity, respiratory muscle strength and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cystic fibrosis
* 8-18 years
* Clinically stable during last six weeks

Exclusion Criteria:

* hemoptysis
* low saturation (SpO2<90%)
* acute lower respiratory tract infection
* cardiac problems (heart failure, arrhythmia, cardiomyopathy, etc.)
* cognitive problems
* pneumothorax

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Cough capacity | 6 weeks
  peak expiratory flow meter

SECONDARY OUTCOMES:
Respiratory muscle strength | every two weeks
  maximal expiratory pressure, maximal inspiratory pressure
Exercise capacity | 6 weeks
  six minute walking test

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Emirza C, Aslan GK, Kilinc AA, Cokugras H. Effect of expiratory muscle training on peak cough flow in children and adolescents with cystic fibrosis: A randomized controlled trial. Pediatr Pulmonol. 2021 May;56(5):939-947. doi: 10.1002/ppul.25259. Epub 2021 Jan 26. PMID 33421333
- [Derived] Stanford G, Ryan H, Solis-Moya A. Respiratory muscle training for cystic fibrosis. Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD006112. doi: 10.1002/14651858.CD006112.pub5. PMID 33331663
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/23143864